CLINICAL TRIAL: NCT00069303
Title: Investigation of the Natural History of West Nile Virus Infection in Patients With Recently Acquired West Nile Fever or Neuroinvasive Disease
Brief Title: Natural History of West Nile Virus Infection
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030305; 03-CC-0305
Record Dates: First submitted 2003-09-22; First posted 2003-09-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-18

CONDITIONS: West Nile Virus; Encephalitis; Myelitis
Keywords: West Nile Virus; Encephalitis; Virus; Mosquito; Fever; WNV; Myelitis
MeSH Terms: conditions — Encephalitis; Myelitis; Virus Diseases; Fever

SUMMARY:
This study will examine how West Nile virus (WNV) infection affects the body. Some people infected with WNV have no symptoms. In others, symptoms may vary from fever and headache to a polio-like syndrome with paralysis, to coma and brain changes like those of a stroke. Many patients recover with no lasting effects, while a few can have long-lasting neurological damage or may die. This study will collect clinical, laboratory, diagnostic, and radiographic information on people thought to have WNV to better understand the disease.

Patients 18 years of age and older diagnosed with or suspected of having West Nile virus infection may be eligible for this study. Patients will be hospitalized until they are well enough to go home and will undergo the following tests and procedures:

* Medical history and physical examination: A thorough history and physical examination will be done on the first day of the study. Then, brief physical exams, including measures of blood pressure, heart rate, breathing rate, and temperature, will be done during each day of hospitalization and at every follow-up clinic visit (at 2 weeks and at 1, 3, and 6 months).
* Blood tests: Blood samples will be collected on the first day of the study, at day 7, at hospital discharge, and at follow-up visits to determine if virus remains in the blood and how it is affecting the body.
* Magnetic resonance imaging (MRI): MRI scans will be done within 72 hours of beginning the study and 1 month after that. This test uses a strong magnetic field and radio waves to produce images of the brain that might show abnormalities in the brains of patients with WNV and reveal whether the abnormalities can predict how an individual will recover. For the procedure, the patient lies on a table that is moved into the narrow tunnel-like scanner. During the procedure, a contrast agent that brightens the images is injected through a catheter placed in an arm vein.
* Neurological examination and neurological function tests: Participants will be tested to see if the West Nile virus has affected their thinking and ability to perform normal daily activities. These tests will be done at the start of the study, on days 3 and 7 (also days 2, 4, 5, and 6 if patients are still in the hospital), at discharge, and at follow-up visits. The tests involve answering a number of questions and performing simple tasks, such as squeezing a hand or lifting a foot.
* Patients who develop weakness in their arms or legs will also have the following studies:

  1. Electromyography (EMG) to study the electrical activity of the muscle. For this test, needles are placed into a muscle to record the electrical activity at that site.
  2. Nerve conduction studies to measure how well the nerves are working. A small charge of electricity is delivered to a nerve in the affected limb, triggering a muscle to tighten or bend. Small wire electrodes are attached to the skin to measure the time is takes for the nerve to move the electrical current from one part of the limb to another.
  3. Spinal MRI to see if the virus is affecting the spinal cord.

Results of other tests done by the patient's local doctor (such as lumbar puncture, electroencephalogram, x-rays, etc.) will be requested. If a lumbar puncture is done, a small amount of cerebrospinal fluid will be requested for testing for WNV.

DETAILED DESCRIPTION:
Investigation of the Natural History of West Nile Virus Infection in Patients with Recently Acquired West Nile Fever or Neuroinvasive Disease is a descriptive natural history study. Since the first reports of WNV disease in North America in 1999, geographic range has expanded, a trend that is expected to continue for the near future. There are few sequentially collected clinical, radiologic and laboratory data from patients with WNV disease. Standardized data collection tools to measure neurologic outcome have not been developed. Prospectively collected data on laboratory and clinical events associated with WNV infection are needed to bridge gaps in current knowledge of this disease and to assist with the design of better treatments. The objectives of this study are to identify and describe the mortality and morbidity, specifically the neurologic and functional outcomes of patients with confirmed WNV disease in order to characterize the clinical course and diverse manifestations, and to assess kinetics of humoral immune responses to WNV infection, correlating these responses with clinical outcomes. Eligible patients fall into two categories: those with neuroinvasive disease caused by WNV infection, and those with WNV fever who received medical attention for their illness. All subjects must have had illness onset within four months prior to enrollment and must have laboratory confirmation of the diagnosis. There will be study visits at Days 1, 14, 30, 90, 180, and 365. Evaluations will include serum and cerebrospinal fluid for determination of WNV IgM/IgG levels and PCR for WNV, urine PCR for WNV, physical examination, serial neurologic examinations, a baseline MRI scan, and four functional and cognitive assessments that have been validated in neurologic illness in adults: the Barthel Index (BI), the Modified Rankin Scale (MRS), the Glasgow Outcome Score (GOS) and the modified Mini-Mental Status Examination (3MS). The subset of study participants who develop motor weakness of an extremity (ies) will have electromyograms, nerve conduction studies and spinal MRI performed. Results from selected clinically indicated tests (done by study participants' physicians, not mandated for the study) will be recorded in the Case Record Forms (CRFs).

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients, regardless of race or gender, who consent and meet entry criteria will be enrolled, according to the following criteria. Note: Due to the low case incidence and the lack of validation of the neurologic scoring systems in children, enrollment will be restricted to adults. Two cohorts of patients will be enrolled: Neuroinvasive Disease and West Nile Fever.

Greater than or equal to 18 years of age.

Documented WNV infection (fever or neuroinvasive disease) that began within four months prior to study entry. Illnesss onset is defined as the first visit to a medical care provider where compatible symptoms (see cohort A or B below) are documented.

Local laboratory documentation of WNV infection as defined by positive IgM and/or PCR for WNV in serum or CSF concurrent with or following illness onset.

Qualification for Cohort A or B:

A. Neuroinvasive Disease Cohort:

- Fever (temperature greater than 38 C) documented by a health care provider

AND: at least one of the following, as documented by a health care provider and in the absence of a more likely clinical explanation:

* Acutely altered mental status (e.g., disorientation, obtundation, stupor, or coma),
* Other acute signs of central or peripheral neurologic dysfunction (e.g., paresis or paralysis, nerve palsies, sensory deficits, abnormal reflexes, generalized convulsions, or abnormal movements), or
* Cerebrospinal fluid (CSF) pleocytosis (white blood cell count greater than or equal to 4 per mm(3) corrected for red blood cell contamination in CSF) associated with illness clinically compatible with meningitis (e.g., headache or stiff neck)

B. West Nile Fever Cohort:

- Temperature greater than 38 C as documented by a health care provider.

EXCLUSION CRITERIA:

Unable to obtain valid informed consent.

Alternate explanation (as determined by the investigator) for clinical findings (such as structural brain lesion, cerebrovascular accident, or other infectious disease).

Evidence of a microbial organism demonstrable on gram or fungal stain of CSF within four months prior to study entry.

Investigator's opinion that patient would be unable to adhere to protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2003-09-16; Study Completion 2011-02-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mostashari F, Bunning ML, Kitsutani PT, Singer DA, Nash D, Cooper MJ, Katz N, Liljebjelke KA, Biggerstaff BJ, Fine AD, Layton MC, Mullin SM, Johnson AJ, Martin DA, Hayes EB, Campbell GL. Epidemic West Nile encephalitis, New York, 1999: results of a household-based seroepidemiological survey. Lancet. 2001 Jul 28;358(9278):261-4. doi: 10.1016/S0140-6736(01)05480-0. PMID 11498211
- [Background] Nash D, Mostashari F, Fine A, Miller J, O'Leary D, Murray K, Huang A, Rosenberg A, Greenberg A, Sherman M, Wong S, Layton M; 1999 West Nile Outbreak Response Working Group. The outbreak of West Nile virus infection in the New York City area in 1999. N Engl J Med. 2001 Jun 14;344(24):1807-14. doi: 10.1056/NEJM200106143442401. PMID 11407341
- [Background] Kelley TW, Prayson RA, Isada CM. Spinal cord disease in West Nile virus infection. N Engl J Med. 2003 Feb 6;348(6):564-6; author reply 564-6. doi: 10.1056/NEJM200302063480618. No abstract available. PMID 12571269